CLINICAL TRIAL: NCT05647369
Title: The Effect of Chios Mastic Mouthwash on Halitosis and Oral Hygiene in Orthodontic Patients: a Randomized Clinical Trial
Brief Title: Chios Mastic Mouthwash and Halitosis and Oral Hygiene in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iosif Sifakakis (Other)
Responsible Party: Sponsor-Investigator, Iosif Sifakakis, Iosif Sifakakis, assistant professor, National and Kapodistrian University of Athens, University of Athens
Organization: University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 461/12.03.2021
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Halitosis; Orthodontic Appliance Complication
Keywords: Halitosis; Mastic; Orthodontic appliance
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Intervention Model Description: This trial is designed as a prospective, randomized, placebo-controlled, double (investigator and patient) blinded, with two parallel groups and an equal allocation ratio in all groups. In this study, the intervention consists of delivery of mastic mouthwash or placebo lozenges.
Who Masked: Participant, Investigator
Masking Description: All patients will be allocated at a 1:1 ratio between group A (mastic group) and group B (placebo group), for each sex separately using stratified randomization. Two random sequences of 15 letters (A or B) will be obtained from www.random.org (List Randomizer service), one for males and one for females. Those letters were written on paper and then sealed in opaque envelopes, sequentially numbered from M1 to M15 for males and from F1 to F15 for females respectively. All envelopes were sealed, numbered and stored in a drawer by a person not involved in the study. Every patient enrolled in the study will receive an envelope in a numerical order and their name was written on the envelope. Informed consent will be obtained from parents / legal guardians and written consent upon information and prior to the randomization or application of any procedure obtained from the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Group 1 (Experimental): Experimental: Experimental group 1: patients, age 13-18, conventional brackets, Mastic mouthwash 15 patients, age 13-18,with conventional brackets,will get Mastic mouthwash
  Interventions: Dietary Supplement: Mastic mouthwash
- Control group: Group 2 (Placebo Comparator): Control group: Group 2 patients, age 13-18, conventional brackets, placebo mouthwash 15 patients, age 13-18,with conventional brackets,will get placebo mouthwash
  Interventions: Dietary Supplement: Placebo mouthwash

INTERVENTIONS:
Dietary Supplement: Mastic mouthwash — All 30 patients will be randomly assigned to either the mastic mouthwash group A (Art of Nature Mastiha Mouthwash, Mastihashop, Greece) (n = 15) or the placebo mouthwash group B (from the same manufacturer) (n = 15) (Table 1). All patients will be asked to use the mouthwash twice a day (10 ml of mouthwash / 2 times a day for 30 sec for 14 days, every morning and every night after brushing) and to maintain their usual oral hygiene routine. The measurements will be done in the morning and at least three hours after brushing and without the use of the mouthwash by the participant on the day of the assessments.
  Arms: Experimental: Group 1
Dietary Supplement: Placebo mouthwash — All 30 patients will be randomly assigned to either the mastic mouthwash group A (Art of Nature Mastiha Mouthwash, Mastihashop, Greece) (n = 15) or the placebo mouthwash group B (from the same manufacturer) (n = 15) (Table 1). All patients will be asked to use the mouthwash twice a day (10 ml of mouthwash / 2 times a day for 30 sec for 14 days, every morning and every night after brushing) and to maintain their usual oral hygiene routine. The measurements will be done in the morning and at least three hours after brushing and without the use of the mouthwash by the participant on the day of the assessments.
  Arms: Control group: Group 2

SUMMARY:
Halitosis is the third most common oral condition perceived by the patients as pathologic, after caries and periodontal diseases. Although it is difficult to estimate the prevalence of halitosis in the population due to the different assessment methods, the available descriptive epidemiologic studies estimate that 30-50% of the population experience oral malodor. Pathologic halitosis most commonly (85%) originates from the oral cavity and is a result of bacterial deposits that cover the tongue or are found in the inflamed oral mucosa, under poor-quality restorations, orthodontic mechanisms, carious lesions or mucosal ulcers. Odor usually results from the microbial degradation of organic substrates present in saliva. This interaction generates malodorous volatile sulfur compounds (VSCs), of which the three most common are: hydrogen sulfide (H2S), methyl-mercaptan (CH3SH) and dimethyl sulfide [(CH3)2S].

Orthodontic patients with fixed appliances are more prone to halitosis, due to the increased plaque accumulation and the increased amounts of available nutrients for the supragingival and subgingival microbes .

DETAILED DESCRIPTION:
AIM: The aim of this study is to investigate the effect of Mastic mouthwash on halitosis (Volatile Sulfur Compounds' levels, VSCs) as well as plaque and gingival indexes in patients undergoing orthodontic treatment with fixed appliances PARTICIPANTS AND METHOD: The study is a double-blinded, placebo-controlled, parallel group, randomized clinical trial. Thirty patients with fixed orthodontic appliances were randomly allocated at a 1:1 ratio, to either the mastic-mouthwash or the placebo-mouthwash group. Eligibility criteria included ages between 13 and 18, active orthodontic treatment with fixed appliances, good general health and total initial VSCs levels above the baseline level of 150ppb. The primary outcomes will be: (a) their subjective perception of their own malodor via questionnaires, (b) their objective VSCs levels (hydrogen sulfide (H2S), methyl-mercaptan (CH3SH) and dimethyl sulfide ((CH3)2S) through the OralChromaTM device and (c) oral hygiene assessed with the use of the Modified Silness and Löe Plaque Index (PI-M) and the Silness and Löe Gingival Index (GI). Measurements were taken at baseline (T0) and after 2 weeks (T1).

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for the trial must comply with all of the following at randomization:

• Age between 13 and 18 years for the group with conventional orthodontic appliances.

This age group represents the majority of patients seeking orthodontic treatment and is homogeneous regarding occupational status (high-school and lyceum students in Greece). Younger patients might present with cooperation problems.

* Good general health.
* Orthodontic fixed labial appliances on the maxillary and mandibular arch, brackets at least on 20 teeth for more than 4 months before enrollment and estimated duration of the treatment more than 1 month, bands on the first molars, extraction cases patients could be enrolled at least two months after the last extraction.
* Total initial VSCs levels above the baseline level of 150ppb.

Exclusion Criteria:

Patients will be excluded for any of the following reasons:

* Active caries
* Periodontitis
* Dental fluorosis / dysplasia of the teeth
* Syndromes, mental disabilities and craniofacial deformities
* Smoking or use of other tobacco products
* Allergy to mastic
* Antibiotics during the last 2 months
* Chlorhexidine in the previous 3 weeks
* Participation in other trials

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Modified plaque index (PI-M) | baseline-2 weeks
  The Silness and Löe index (Silness and Löe, 1964) does not take into account the pattern of plaque accumulation in orthodontic patients. To overcome this problem, Williams et al. (1991) divided the tooth into mesial, distal, gingival, and incisal regions in relation to the bracket and scored plaque in each region using the four codes of the original index (0 to 3). The values are summed to obtain a total score, which ranges from 0 to 12 for each tooth. This modified index is recommended for patients with fixed orthodontic appliances because it acknowledges the usual effects of orthodontic appliances on plaque distribution and has much greater categorical discrimination.
Gingival index (GI) | baseline-2 weeks
  The Gingival Index (GI) is a measure of the severity of gingivitis and is scored by measuring the amount of gingival inflammation, also considering redness and bleeding (Löe & Silness, 1963).
VSCs levels {hydrogen sulfide (H2S), methyl-mercaptan (CH3SH) and dimethyl sulfide [(CH3)2S]. | baseline-2 weeks
  VSCs levels {hydrogen sulfide (H2S), methyl-mercaptan (CH3SH) and dimethyl sulfide [(CH3)2S]} will be measured with the OralChromaTM device (NOVATRONIC Deutschland GmbH, Kölner Straße 102, D-51429 Bertogisch Gladbach).
  The organoleptic evaluation will be done by the patient, due to the current pandemic of the SARS-Covid 19 virus. This assessment will be subjectively based on a scale in printed questionnaires. The objective assessment of the T0-T1 VSCs levels will be done with the OralChromaTM. This chromatograph measured the concentrations of the oral gases H2S, CH3SH and (CH3)2S. The sample will be collected using disposable syringes (1 ml plastic syringes), which will be inserted into the patient's oral cavity. The patients weill be asked to close their mouth for 30 seconds before the samples collection. Then 0.5ml of air will injected from the syringe's intake into the measuring device.

CONTACTS AND LOCATIONS:
Overall Officials: Iosif Sifakakis, Assistant Professor, Principal Investigator — University of Athens
Locations (1):
- National and Kapodistrian University of Athens, School of Dentistry, Departments of Orthodontics, Athens, Attica, Greece

REFERENCES:
- [Derived] Tsironi K, Mylonopoulou IM, Pandis N, Vassilopoulos S, Sifakakis I, Papaioannou W. The effect of mastic mouthwash on halitosis and oral hygiene in orthodontic patients: a randomized clinical trial. Eur J Orthod. 2023 Nov 30;45(6):781-787. doi: 10.1093/ejo/cjad036. PMID 37503575